CLINICAL TRIAL: NCT06374017
Title: Evaluating the Effect of Topical Lidocaine Spray Versus Dexmedetomidine Spray on Suppression of Stress Response to Laryngoscopy and Endotracheal Intubation: a Randomized Controlled Study
Brief Title: Evaluation of Lidocaine Spray Versus Dexmetomidine Spray on Stress Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Mohamed, Lecturer of Anesthesia and Surgical ICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-258-2023
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: To Measure Systolic Blood Pressure Postintubation
MeSH Terms: interventions — Saline Solution; Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): Group C: will receive 5ml of normal saline sprayed via long nostril syringe into oropharynx, the vocal cords and tracheobronchial tree 5 minutes before intubation
  Interventions: Drug: Normal saline, Lidocaine, dexmetomidine
- Group L (Active Comparator): : : will receive 5ml of lidocaine 2% (100mg) sprayed via long nostril syringe into oropharynx , the vocal cords and tracheobronchial tree 5 minutes before intubation
  Interventions: Drug: Normal saline, Lidocaine, dexmetomidine
- Group D (Active Comparator): will receive dexmedetomidine (1 μg/kg) diluted in 5ml normal saline sprayed via long nostril syringe into oropharynx , the vocal cords and tracheobronchial tree 5 minutes before intubation.
  Interventions: Drug: Normal saline, Lidocaine, dexmetomidine

INTERVENTIONS:
Drug: Normal saline, Lidocaine, dexmetomidine — The study drug of each group will be sprayed into oropharynx, the vocal cords and tracheal tree 3 minutes after induction of anesthesia and 5 minutes before intubation.

SUMMARY:
Many studies discussed attenuating stress response by various measures but to the interest of our study , No one compared topical spray of both lidocaine and dexmedetomidine in attenuating the haemodynamic stress responses of laryngoscopy and endotracheal intubation, avoiding undesired systemic effects of drugs ,

DETAILED DESCRIPTION:
This study will be conducted in the operating theatres of Cairo university hospitals.

Patients undergoing any surgery under general anesthesia and needs endotracheal intubation using direct laryngoscopy will be assigned to one of the three groups:

Group C: will receive 5ml of normal saline sprayed via long nostril syringe into oropharynx, the vocal cords and tracheobronchial tree 5 minutes before intubation Group L: : will receive 5ml of lidocaine 2% (100mg) sprayed via long nostril syringe into oropharynx , the vocal cords and tracheobronchial tree 5 minutes before intubation Group D: : will receive dexmedetomidine (1 μg/kg) diluted in 5ml normal saline sprayed via long nostril syringe into oropharynx , the vocal cords and tracheobronchial tree 5 minutes before intubation.

ELIGIBILITY:
Inclusion Criteria:

* • ASA I,II

  * Age 18-60y
  * Patients scheduled for any operations under general anesthesia and needs endotracheal intubation using direct laryngoscopy in the operating theatre.

Exclusion Criteria:

* • Uncontrolled high blood pressure > 160/100 heart disease in the form of ischemic heart disease and severe valvular disease.

  * Patients with the history of allergy to lidocaine or dexmedetomidine.
  * ASA III & IV.
  * Patients refuse to share in this study
  * Suspected difficult intubation that needs more than 2 trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
To measure systolic blood pressure immediately after intubation. | Immediately after endotracheal intubation
  Using invasive blood pressure monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospitals, Cairo, Egypt